CLINICAL TRIAL: NCT04350957
Title: Low-dose Imaging Technique (LITE) MRI Gadavist® (Gadobutrol)
Brief Title: Low-dose Imaging Technique (LITE)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution due to family emergency prior to IRB approval.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB20-0528
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: This clinical trial has a single arm. All subjects will receive a low dose and standard dose on two separate days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low-dose Imaging (Experimental): Enrolled patients will undergo two separate dynamic contrast-enhanced MRI's, one with 25% of the contrast dose and one with 100% of the contrast dose recommended by weight. During the first visit, the subject will receive 25% of the standard dose of contrast media 0.1 mM/kg will be administered at 2 mls/second followed by the acquisition of a series of DCE images. On the second visit, the subject will receive 100% of the contrast media followed by the same imaging protocol as the one subsequent to the first contrast administration.
  Interventions: Diagnostic Test: Low-dose Imaging

INTERVENTIONS:
Diagnostic Test: Low-dose Imaging — We are comparing MRI image quality for diagnostic purposes. We hope to learn whether using a lesser dose (25%) of the FDA approved contrast agent, Gadavist®, is just as effective as a standard or full dose (100%) of the same contrast in a breast MRI.
  This research is being done because breast MRI's have repeatedly been shown to represent the most reliable imaging method for breast cancer screening and diagnosis, regardless of personal risk for breast cancer and radiographic breast density. However, there are growing concerns about getting frequent breast MRI examinations due to the deposition of gadolinium, a metal ion that is found in all breast MRI contrast agents. The FDA states that this deposition and retention is not known to have any long term side effects on patient. However, the researchers at the University of Chicago Medicine would like to further investigate this using a lesser dose of contrast agent than the recommended dose for breast MRI examinations.

SUMMARY:
The purpose of this study is to compare the diagnostic accuracy of a breast MRI when using a smaller dose of contrast compared to a full dose of contrast.

Each patient will be injected with a low-dose and standard dose of Gadavist® acquired on two separate days. Both low-dose and standard-dose images for each patient will allow matched comparison for comprehensive quantitative evaluation. To evaluate these diagnostic methods we need volunteers who are willing to allow us to take a number of different MRI pictures of their breasts. The scans we are asking you to volunteer for now is for research purposes only and will have no effect on the medical care you receive from your doctors.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-80
* Women with a suspected or biopsy proven enhancing lesion

Exclusion Criteria:

* Women with a history of adverse reactions to contrast media
* Women with GFR below 30 mL/min/1.73m2
* Women who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Low-dose Lesion Enhancement | Through study completion, an average of 1 year
  Readers will initially be provided with two MIP images and asked to decide on presence or absence of significant enhancement. The two MIP images will be created from the low dose images and the standard dose images respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Sheth, MD, Principal Investigator — University of Chicago; Gregory S Karczmar, PhD, Principal Investigator — University of Chicago